CLINICAL TRIAL: NCT00820820
Title: Immunotherapy of Atopic Dermatitis in Adult Patients by Anti-measles Vaccination IDA (Immunothérapie de la Dermatite Atopique)Protocol
Brief Title: IDA (Immunothérapie de la Dermatite Atopique) Adult - Immunotherapy in Atopic Dermatitis
Acronym: IDA-Adult
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: C07-38; 2007-007267-25 (EudraCT Number)
Record Dates: First submitted 2009-01-09; First posted 2009-01-12 (Estimated); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Atopic Dermatitis
Keywords: Atopic Dermatitis; immunosuppression; Measles vaccine; T lymphocytes; Atopic Dermatitis in adults
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rouvax (Active Comparator)
  Interventions: Biological: ROUVAX
- Placebo (Placebo Comparator): Sub cutaneous injection of vehicle
  Interventions: Biological: placebo

INTERVENTIONS:
Biological: ROUVAX — Measles vaccine (ROUVAX ®), Schwarz strain (>1000 DICC 50) in 0.5 ml of water for injection. One single subcutaneous injection.
  Arms: Rouvax
Biological: placebo — Vehicle (water for injection), 0.5 ml, once
  Arms: Placebo

SUMMARY:
Atopic dermatitis (AD) is a chronic inflammatory disease of the skin. AD is very frequent, and involves T lymphocytes cells. Measles vaccination, as well as measles vaccine, induces a temporary immunosuppression; furthermore, an improvement of AD has been observed during measles infection.

This trial is aimed at demonstrating that measles vaccine is able to create an immunomodulation and to improve AD symptoms.

30 adult patients of both sexes with moderate to severe AD will be randomly assigned to measles vaccine (ROUVAX ®), or placebo (vehicle) and follow-up for 45 days.

The primary outcome is the effect of anti-measles vaccination on the T cell responses in patients; Other outcomes include: clinical evolution of AD, as measured by the SCORAD, the evolution of blood level of measles specific IgE and antibodies; evolution of other biomarkers and phenotypic characteristics of T lymphocytes.

DETAILED DESCRIPTION:
Atopic dermatitis (AD) is a chronic inflammatory disease of the skin. AD is very frequent, and involves T lymphocytes cells. Measles vaccination, as well as measles vaccine, induces a temporary immunosuppression; furthermore, an improvement of AD has been observed during measles infection.

This trial is aimed at demonstrating that measles vaccine is able to create an immunomodulation and to improve AD symptoms.

ELIGIBILITY:
Inclusion Criteria:

* adults patients of both sexes, with moderate to severe Atopic Dermatitis (SCORAD (Score for Atopic Dermatitis) ≥ 15).

Exclusion Criteria:

* hypersensititvity or contra-indication to a Rouvax® component, Tubertest® component, to egg proteins, immunological deficiency, pregnancy, neomycin
* allergy,
* systemic immnosuppressive treatment in the previous 3 months,
* topic immunosuppressive treatment during the week preceeding the inclusion (gluco-corticoid, or immunosuppressive agent),
* fever or acute disease (the inclusion must be postpone in such cases).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-01-09 (Actual); Primary Completion 2012-03-26 (Actual); Study Completion 2012-03-26 (Actual)

PRIMARY OUTCOMES:
Effect of anti-measles vaccination on the T cell responses in patients | 7 / 10 days after vaccine / placebo injection

SECONDARY OUTCOMES:
Clinical evolution of AD, as measured by the SCORAD | 3 weeks after injection
blood level of measles specific IgE and antibodies | 3 weeks after injection
Biomarkers - E selectin, CD25, soluble CD30, CCL 17 and CCL 18 | 7 days, 14 days, 3 weeks after injection
phenotypic characteristics of T lymphocytes | 7 days, 14 days, 3 weeks, and 6 weeks after injection

CONTACTS AND LOCATIONS:
Overall Officials: Branka Horvat, MD, PhD, Study Director — Institut National de la Santé Et de la Recherche Médicale, France
Locations (1):
- Unité de Recherche Clinique et Immunologique, Pierre-Bénite, Lyon, France